CLINICAL TRIAL: NCT00906074
Title: A Multicenter, Surgeon-Matched Case-Control Study of Severe Surgical Site Infections (SSIs) Following Contaminated Or Dirty-infected Abdominal Surgery
Brief Title: Study Evaluating Severe Surgical Site Infections (SSIs) Following Contaminated Or Dirty-infected Abdominal Surgery
Acronym: EURIDICE
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1811046; 3074A1-4463 (Other: Wyeth)
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Results first posted 2012-04-11 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Surgical Wound Infection; Postoperative Wound Infection
Keywords: Surgical Wound Infection; Surgical Site Infection; Abdominal Surgery
MeSH Terms: conditions — Surgical Wound Infection | interventions — Elective Surgical Procedures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case: Cases will be defined as patients with elective or emergency abdominal surgery who develop severe surgical site infection (deep incisional or organ cavity type; see Center for Disease Control (CDC) criteria for definition in the Appendix), within 0-30 days of surgery.
  Interventions: Procedure: Elective or emergency abdominal surgery
- Control: Surgeon-matched controls will be patients with elective or emergency abdominal surgery who are free of surgical site infection (SSI) after 30 days from the surgery.
  Interventions: Procedure: Elective or emergency abdominal surgery

INTERVENTIONS:
Procedure: Elective or emergency abdominal surgery — Clinical record review.
  Groups: Case
Procedure: Elective or emergency abdominal surgery — Clinical record review
  Groups: Control

SUMMARY:
This is an observational study to evaluate the relative importance of the known risk factors for severe surgical site infections (SSIs) on the development of the more severe SSI cases, and to describe the demographic, clinical features, etiology and the management and outcome of patients suffering from severe SSIs in Spain.

DETAILED DESCRIPTION:
Case and Control study.

ELIGIBILITY:
Inclusion Criteria:

* Age of or above 18 years.
* Admitted to a General Surgery Ward for elective or emergency abdominal surgery.
* Contaminated or dirty-infected surgical procedures.
* Only for cases, they will have to present symptoms and signs of a surgical site infection (SSI) (within 0-30 days) after abdominal surgery.
* Only for controls, patients must be free of SSI after 30 days from surgery, regardless of whether they are still in the hospital or being observed as an outpatient in the external clinic.

Exclusion Criteria:

* Age under 18 years.
* American Society of Anesthesiologist (ASA) score of 5 or above.
* Surgical implant in place.
* Clean or clean-contaminated surgical procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with or without surgical site infections (SSI) after surgery, treated in major hospitals with general surgical units selected from all over Spain
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2009-02; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1811046&StudyName=Study%20Evaluating%20Severe%20Surgical%20Site%20Infections%20%28SSIs%29%20Following%20Contaminated%20Or%20Dirty-infected%20Abdominal%20Surgery

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 289 participants were screened and 109 were excluded from analysis due to: no matching control, not meeting inclusion/exclusion criteria or did not meet matching criteria.
Groups:
- Case: Cases were defined as participants with severe surgical site infection (SSI) (deep incisional or organ space type; see Center for Disease Control [CDC] criteria for definition in the Appendix) in participants who underwent elective or emergency abdominal surgery in the previous 30 days.
- Control: Participants who were free of surgical site infection (SSI) within 30 days following surgeon matched elective or emergency abdominal surgery.
Period: Overall Study
Arm/Group | Case | Control
Started | 90 | 90
Completed | 90 | 90
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Case | Control | Total
Number analyzed (Participants) | 90 | 90 | 180
Age Continuous [Mean (Standard Deviation); unit: years] | 62.49 (16.11) | 58.46 (20.40) | 60.47 (18.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 39 | 66
  Male | 63 | 51 | 114

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Pre-surgical Morbidities
Description: Morbidities (risk factors) included: neoplasm, tobacco use, body mass index (weight in kilograms divided by height in meters squared [BMI kg/m2]) greater than (>) 30, diabetes mellitus (DM), immunosuppression/ corticosteroids, anemia (hemoglobin [Hb] less than (>) 9 grams per deciliter [gr/dL]) or malnutrition (hypoalbuminemia).
Time Frame: Baseline (Pre-surgical)
Population: Study population: participants with or without SSI after surgery, treated in major hospitals with general surgical units located in Spain
Measure: Number; unit: percentage of participants
Arm/Group | Case | Control
Number analyzed (Participants) | 90 | 90
percentage of participants
  Neoplasm | 47.8 | 48.9
  Tobacco use | 26.7 | 23.3
  BMI kg/mˆ2>30 | 23.3 | 12.2
  Diabetes mellitus | 17.8 | 11.1
  Immunosuppression/corticosteroids | 7.8 | 7.8
  Anemia (Hb<9 gr/dL) | 7.8 | 2.2
  Malnutrition (hypoalbuminemia) | 4.4 | 2.2
Statistical Analysis 1: Comparison: Case vs Control; Neoplasm; Test type: Superiority or Other; p = 0.881, Chi-squared; Chi-squared Pearson
Statistical Analysis 2: Comparison: Case vs Control; Tobacco use; Test type: Superiority or Other; p = 0.517, Chi-squared; Chi-squared Pearson
Statistical Analysis 3: Comparison: Case vs Control; BMI(kg/mˆ2)>30; Test type: Superiority or Other; p = 0.053, Chi-squared; Chi-squared Pearson
Statistical Analysis 4: Comparison: Case vs Control; Diabetes mellitus; Test type: Superiority or Other; p = 0.289, Chi-squared; Chi-squared Pearson
Statistical Analysis 5: Comparison: Case vs Control; Immunosuppression/Corticosteroids; Test type: Superiority or Other; p = 1.000, Chi-squared; Chi-squared Pearson
Statistical Analysis 6: Comparison: Case vs Control; Anemia (Hb<9gr/dL); Test type: Superiority or Other; p = 0.169, Chi-squared; Chi-squared Pearson
Statistical Analysis 7: Comparison: Case vs Control; Malnutrition (hypoalbuminemia); Test type: Superiority or Other; p = 0.637, Chi-squared; Chi-squared Pearson

2. Primary Outcome: Percentage of Participants Who Received Pre-surgical Antibiotic Prophylaxis
Time Frame: Baseline (Pre-surgical)
Population: Study Population
Measure: Number; unit: Percentage of participants
Arm/Group | Case | Control
Number analyzed (Participants) | 90 | 90
Percentage of participants | 95.5 | 96.7
Statistical Analysis 1: Comparison: Case vs Control; Test type: Superiority or Other; p = 1.000, Chi-squared; Chi-squared Pearson

3. Primary Outcome: Percentage of Participants Who Underwent Emergency Surgery or Scheduled Surgery
Time Frame: Day 0 (day of surgery)
Population: Study Population
Measure: Number; unit: Percentage of participants
Arm/Group | Case | Control
Number analyzed (Participants) | 90 | 90
Percentage of participants
  Emergency surgery | 32.2 | 31.1
  Scheduled surgery | 67.8 | 68.9
Statistical Analysis 1: Comparison: Case vs Control; Test type: Superiority or Other; p = 0.873, Chi-squared; Chi-squared Pearson

4. Primary Outcome: Percentage of Participants With Classification of Risk of Surgical Infection of Clean-contaminated, Contaminated or Dirty
Description: Surgical infection risk class: Clean-contaminated: controlled entry in normally colonized body cavities/no unusual contamination/minimum fluid discharge/minimal sterile technique violation/re-surgery on clean surgical incision within 7 days/negative surgical exploration through intact skin. Contaminated: no acute inflammation/purulent discharge/significant fluid/material violation of sterile technique/penetrating trauma less than 4 hours old/graft in chronic skin wounds. Dirty: pus-abscess drainage/ preoperatively colonized body cavity perforated/penetrating trauma more than 4 hours old.
Time Frame: Day 0 (day of surgery)
Population: Study population
Measure: Number; unit: Percentage of participants
Arm/Group | Case | Control
Number analyzed (Participants) | 90 | 90
Percentage of participants
  Clean-contaminated | 60.0 | 60.0
  Contaminated | 30.0 | 30.0
  Dirty | 10.0 | 10.0

5. Primary Outcome: Type of Surgeon
Description: Surgical speciality of physician who performed surgery.
Time Frame: Day 0 (day of surgery)
Population: No data collected
Measure: Number; unit: surgeon
Arm/Group | Case | Control
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Percentage of Participants With Infection
Description: Microorganism infection by bacterial type.
Time Frame: Day 0 (day of surgery) up to 30 days post surgery
Population: Subset of study population with infection; N=number of participants with evaluable data
Measure: Number; unit: Percentage of participants
Arm/Group | Case
Number analyzed (Participants) | 86
Percentage of participants
  Escherichia coli (E. coli) | 55.8
  Bacteroides fragilis group (gr.) | 14.0
  Enterococcus faecium | 12.8
  Enterococcus faecalis | 12.8
  Pseudomonas aeruginosa | 8.1
  Staphylococcus epidermidis | 7.0
  Candida albicans | 5.8
  Staphylococcus species (spp) | 5.8
  Morganella morganni | 5.8
  Klebsiella oxytoca | 5.8
  Klebsiella pneumoniae | 4.7
  Streptococcus spp | 3.5
  Streptococcus other | 3.5
  Streptococcus anginosus | 3.5
  Staphylococcus aureus | 3.5
  Extended-spectrum β-lactamase producing E.coli | 3.5
  Enterobacter cloacae | 3.5
  Streptococcus viridians gr. | 2.3
  Streptococcus agalactiae | 2.3
  Coagulase-negative staphylococci | 2.3
  Serratia marcescens | 2.3
  Prevotella spp | 2.3
  Enterococcus spp | 2.3
  Enterococcus durans | 2.3
  Bacteroides vulgates bacteroides (B) fragilis gr. | 2.3
  Candida glabrata | 1.2
  Stenothropomonas maltophilia | 1.2
  Methicillin-resistant Staphylococcus aureus | 1.2
  Serratia spp | 1.2
  Pseudomonas stutzeri | 1.2
  Proteus vulgaris | 1.2
  Lactobacillus spp | 1.2
  Haemophilus parainfluenzae | 1.2
  Gemella spp | 1.2
  Eubacterium gr. | 1.2
  Enterococcus avium | 1.2
  Enterobacter agglomerans | 1.2
  Citrobacter freundii | 1.2
  Bacteroides no fragilis gr. | 1.2
  Bacteroides thetaiotaomicrom B. fragilis gr. | 1.2
  Bacteroides ovatus B. fragilis gr. | 1.2
  Bacteroides distasonis B. fragilis gr. | 1.2
  Non-fermenting gram negative bacilli | 1.2

7. Primary Outcome: Percentage of Participants Who Showed Clinical Improvement of SSI
Description: Clinical improvement of SSI was defined as healed (signs and symptoms of initial infection resolved) or improved (initial signs and symptoms significantly diminished without the appearance of new signs).
Time Frame: Day 0 (day of surgery) up to 30 days post surgery
Population: Subset of study population with infection; N=number of participants with evaluable data
Measure: Number; unit: Percentage of participants
Arm/Group | Case
Number analyzed (Participants) | 89
Percentage of participants
  healed | 70.8
  Improvement | 27.0

8. Primary Outcome: Percentage of Participants With Post-surgical Drainage
Time Frame: Day 0 (day of surgery) up to 30 days post surgery
Population: Study Population
Measure: Number; unit: Percentage of participants
Arm/Group | Case | Control
Number analyzed (Participants) | 90 | 90
Percentage of participants | 71.1 | 61.1
Statistical Analysis 1: Comparison: Case vs Control; Test type: Superiority or Other; p = 0.156, Chi-squared; Chi-squared Pearson

9. Secondary Outcome: Percentage of Participants Whose National Nosocomial Infection Surveillance System (NNISS) Scores of Preoperative Risk of Infection Were Greater Than >0
Description: Percentage of participants with NNISS score for increased preoperative risk of infection.
Time Frame: Baseline (pre-surgical)
Population: Study population
Measure: Number; unit: Percentage of participants
Arm/Group | Case | Control
Number analyzed (Participants) | 90 | 90
Percentage of participants
  1.5 % increased risk | 23.3 | 26.7
  2.9% increased risk | 50.0 | 56.7
  6.8% increased risk | 23.3 | 14.4
  13.0% increased risk | 3.3 | 2.2
Statistical Analysis 1: Comparison: Case vs Control; Test type: Superiority or Other; p = 0.444, Fisher Exact

10. Secondary Outcome: ASEPSIS Classification in Participants With Serious SSI
Description: Additional treatment, Serous discharge, Erythema, Purulent exudate, Separation of deep tissue, Isolation of bacteria, Stay in hospital prolonged over 14 days (ASEPSIS). ASEPSIS classification is a numerical indication of wound healing progress: satisfactory healing (0-10), disturbance of healing (11-20), minor wound infection (20-30), moderate wound infection (30-40), and severe wound infection (over 40).
Time Frame: Up to 30 days post surgery
Population: Subset of study population with infection
Measure: Number; unit: participants
Arm/Group | Case
Number analyzed (Participants) | 90
participants
  Satisfactory healing | 1
  Disturbance of healing | 12
  Minor wound infection | 58
  Moderate wound infection | 15
  Severe wound infection | 4

11. Secondary Outcome: Classification of SSI Infection
Description: Participants with organ-space or deep incisional SSI.
Time Frame: Day 0 (day of surgery) up to 30 days post surgery
Population: Subset of study population with infection; N=number of participants with evaluable data
Measure: Number; unit: participants
Arm/Group | Case
Number analyzed (Participants) | 89
participants
  Organ-space infection | 60
  Deep incisional infection | 29

12. Secondary Outcome: Percentage of Participants Who Had Microbiologic Resolution of SSI (Sensitivity of Microorganisms to Antibiotics)
Description: Resolution of SSI ranged from eradication (infection cured) to persistence (infection continued).
Time Frame: Day 0 (day of surgery) up to 30 days post surgery
Population: Subset of study population with infection; N=number of participants with evaluable data
Measure: Number; unit: Percentage of participants
Arm/Group | Case
Number analyzed (Participants) | 89
Percentage of participants
  Erradication | 29.2
  Presumed erradication | 57.3
  Persistance | 4.5
  Unknown | 9.0

13. Secondary Outcome: Number of Participants With Antimicrobial Resistance
Description: Microbiological resistance reported for microorganisms that were found at a frequency greater (>) than 5 percent (%).
Time Frame: Day 0 (day of surgery) up to 30 days post surgery
Population: Subset of study population with infection; N=number of participants with evaluable data
Measure: Number; unit: Number of participants
Arm/Group | Case
Number analyzed (Participants) | 88
Number of participants
  E. coli-cephalosporins 3rd generation (Cef-3) | 1
  Escherichia coli-carbapenems (Carb) | 0
  Escherichia coli-fluoroquinolones (FQ) | 7
  Bacteroides fragilis gr. (Cef-3) | 0
  Bacteroides fragilis gr. (Carb) | 1
  Bacteroides fragilis gr. (FQ) | 4
  Enterococcus faecium (Cef-3) | 0
  Enterococcus faecium (Carb) | 1
  Enterococcus faecium (FQ) | 0
  Enterococcus faecalis (FQ) | 2
  Pseudomonas aeruginosa (Cef-3) | 1
  Pseudomonas aeruginosa (Carb) | 1
  Pseudomonas aeruginosa (FQ) | 1
  Staphylococus epidermis (FQ) | 4
  Staphylococus spp (FQ) | 4
  Morganella morganni (Cef-3) | 2
  Morganella morganni (Carb) | 0
  Morganella morganni (FQ) | 0
  Enterococcus faecium (enterococcus vancomycin[EV]) | 0
  Enterococcus faecalis (EV) | 0

ADVERSE EVENTS:
Description: No adverse events were collected.
Arm/Group | Case | Control
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Adverse events and serious adverse events were not collected for this epidemiology study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.